CLINICAL TRIAL: NCT06608693
Title: Effect of Different stretchıng Techniques on Balance and Functionality in Children With Diplegic Cerebral Palsy
Brief Title: Effect of Different Stretching Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Uğur Sözlü, Director, Gazi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: (KAEK-118/055)
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy
Keywords: PNF; Static Stretching; Balance; Functionality
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF stretching group (Experimental): PNF and static stretching methods were applied 2 days a week and 6 repetitions in each session for 4 weeks to the hip flexors. In addition to stretching, both of the groups received a routine treatment program consisting of gluteus maximus and quadriceps strengthening, balance, and walking exercises.
  Interventions: Other: PNF stretching
- Static stretching group (Experimental): PNF and static stretching methods were applied 2 days a week and 6 repetitions in each session for 4 weeks to the hip flexors. In addition to stretching, both of the groups received a routine treatment program consisting of gluteus maximus and quadriceps strengthening, balance, and walking exercises.
  Interventions: Other: Static stretching group

INTERVENTIONS:
Other: PNF stretching — Subjects lay supine on a treatment table, holding one knee to the chest and letting the other leg extend freely toward the floor at the end of the table. This protocol was adapted from previous studies. The hip joint was carefully and gradually lowered towards the floor, with the knee flexing at a 90-degree angle until the individual experienced a mild stretching sensation (Visual analog scale:4-6). Then, the subject performed a sub-maximal voluntary isometric contraction by utilizing the flexor muscles for 20 seconds while resisting the applied force exerted by an examiner through the utilization of a hand-held dynamometer (K-Force Muscle Control). The examiner proceeded to passively manipulate the leg to achieve the desired range of motion (ROM), maintaining it for 20 seconds. This process was repeated six times for each limb. The patient rested for 2 minutes before applying the same technique to the other side.
  Arms: PNF stretching group
Other: Static stretching group — While the patient was lying supine, the hip and knee joints on the non-stretch side were kept in 90⸰ flexion. A sandbag was positioned on the side to be stretched, specifically proximal to the patella, in order to induce a moderate sensation of stretching in the patient. Subsequently, a force was exerted in the direction of hip extension for a duration of 30 seconds. Afterward, the patient was instructed to relax. This process was repeated a total of six times, with a designated 20-second rest period between each repetition. The patient took a two-minute rest before the same technique was applied to the other side. There was no specific order on which side to apply the technique.
  Arms: Static stretching group

SUMMARY:
The aim of this study is to investigate the effect of proprioceptive neuromuscular facilitation (PNF) and static stretching techniques on the balance and functional capabilities of children diagnosed with diplegic cerebral palsy (CP).

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of proprioceptive neuromuscular facilitation (PNF) and static stretching techniques on the balance and functional capabilities of children diagnosed with diplegic cerebral palsy (CP). The study consisted of a group of sixteen children, ranging in age from 8 to 16 years, who were diagnosed with bilateral hip flexor contracture and diplegic cerebral palsy. These children were classified according to the Gross Motor Function Classification System (GMFCS) levels I to III. The children were randomly divided into PNF and static stretching groups. Stretching techniques were applied 2 days a week for 4 weeks, with 6 repetitions in each session. The study assessed various parameters, including hip extension range of motion (ROM), muscle tone intensity based on the Modified Ashworth Scale, hip flexor shortness as determined by the Thomas Test, the time up and go (TUG) test, balance using the Pediatric Berg Balance Scale, and functional status evaluated through the Gilette Functional Walking Assessment Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of CP;
* Age ranging from 6 to 18 years;
* No recent administration of Botulinum Toxin to the lower extremity muscles in the last 6 months;
* An IQ score of 70 or above;
* A Gross Motor Function Classification System (GMFCS) value of 1, 2 or 3;
* Presence of hip flexion contracture;
* Willingness to participate in the study

Exclusion Criteria:

* Concomitant diagnoses aside from CP,
* Presenting with muscle tone ratings of 3 or 4 in the hip muscles according to the Modified Ashworth Scale (MAS),
* Who had undergone tendon lengthening surgery to increase hip flexion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2024-09-27 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Hip extension Range of motion in degrees | 3 months
  Hip extension ROM was measured with a digital goniometer while the patient was lying in the prone position, and the knee was flexed.
Thomas test | 3 months
  The degree of hip flexion contracture was determined using the Thomas test while the patient was supine. The opposite hip was passively moved in the flexion direction as much as possible by a second physiotherapist. In the meantime, the degree of hip flexion on the designated side was assessed using a digital goniometer and documented in degrees. This test was repeated 3 times, and the results were averaged.
Timed Up and Go test (TUG) | 3 months
  Functional status was assessed by the Timed Up and Go test (TUG). The time required for the patient to get up from the chair, walk 3 meters, turn around, walk back to the chair, and sit down was calculated in seconds. The test was repeated 3 times, and the data average was recorded.
The Pediatric Berg Balance Scale (PBBS) | 3 months
  The Pediatric Berg Balance Scale (PBBS) was used to evaluate dynamic balance skills in children with CP. The scale comprises 14 items including sitting balance,standing balance, sitting to standing/standing to sitting, transfers, stepping, reaching forward with outstretched arm, reaching the foor, turning, and placing foot on stool items. Each item ranked from 0 to 4. 0 shows inability to perform the instruction, while 4 shows the ability to perform without any difculty. Maximum total score is 56.
Gilette Functional Assessment Questionnaire (FAQ) | 3 months
  Gillette Functional AssessmentQuestionnaire (FAQ) 22-item asks the respondent to 'Please ratehow easy it is for the patient to do the following activities'followed by brief descriptions of 22 locomotor skills the ﬁve-level (minumum:1, maximum:5) Likert response scale used for the 22 skill items was 'easy', 'a little hard', 'very hard', 'can't do at all',and 'too young for activity'.
Age in years | 3 months
  Age of patients will be recorded
Weight in kilograms | 3 months
  Weights of patients will be recorded
Height in meters | 3 months
  Heights of patients will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Selda Başar, Dr, Study Chair — Gazi University
Locations (1):
- Gazi University, Ankara, Emniyet Mahallesi Bandırma Caddesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No